CLINICAL TRIAL: NCT05072379
Title: Examining the Effectiveness of a Mobile App on Self-care for a Colostomy Among Colorectal Cancer Patients and Family Caregivers
Brief Title: Examining the Effectiveness of a Mobile App on Self-care for a Colostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cheng-Hsin General Hospital (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHGH110-(IU)03
Record Dates: First submitted 2021-08-29; First posted 2021-10-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Colostomy
Keywords: m-Health; Colostomy; Anxiety; quality of life
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 1. mobile health app group
  2. control group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile health app group (Experimental): routine care and mobile health app
  Interventions: Device: colostomy self-care app
- control group (No Intervention): routine care

INTERVENTIONS:
Device: colostomy self-care app — The study will use mixed methods as the study design in which content analysis will be used to identify the content suited for the App based on interviews with participants. A systematic research and development process will be utilized to design the text, videos, and images in the App's simulations to provide accurate, consistent, and complete knowledge of the skills needed for colostomy self-care and contending with any potential emergency.
  Arms: Mobile health app group

SUMMARY:
Colorectal cancer has been one of the most common cancers in Taiwan. Using m-Health Apps to improve accessibility of personal health management has received greater attention and recognition. The purpose of this study is to develop a mobile App and understand its effects on improving colorectal cancer participants and their family caregivers' knowledge of colostomy care, anxiety, and quality of life as well as their satisfaction of the App. The study will use mixed methods as the study design in which content analysis will be used to identify the content suited for the App based on interviews with participants. A systematic research and development process will be utilized to design the text, videos, and images in the App's simulations to provide accurate, consistent, and complete knowledge of the skills needed for colostomy self-care and contending with any potential emergency. The results of this study not only will help colorectal participants and their family caregivers increase their knowledge of self-care for their colostomy, reduce anxiety, and improve quality of life, but it will also help the hospital to provide a high-quality and innovative technology for colorectal cancer participant and their family caregivers. Through this App, the quality of interaction and the rapport developed between healthcare professionals and participants will be enhanced, facilitating participant and family caregivers' responses to emergent situations and their endorsements toward the hospital. Ultimately, participants and their families will increase their satisfaction with the care.

DETAILED DESCRIPTION:
In the first stage, a total of 10 pairs of colorectal cancer participants and their main caregivers will be recruited in the hospital to conduct individual interviews to understand the care and learning needs of colorectal cancer participants and their main caregivers, and then use content analysis to analyze the interviews. The result is used as the connotation of a smartphone application to help participants with colorectal cancer stoma and their main caregivers prepare the knowledge and skills needed during care and respond to emergencies that may occur.

In the second stage, patients with colorectal cancer stoma and their main caregivers who have received individual interviews will be invited to trial and provide qualitative feedback after use to facilitate modification and completion of the surface validity test.

In the third stage, 30 pairs of colorectal cancer stoma participants and main caregivers will be recruited in the experimental group and the control group in a randomized controlled design, and the effectiveness of this mobile application will be evaluated by a questionnaire survey before and after the test.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years old
2. The main caregiver for women who are diagnosed with colorectal cancer for the first time and have a stoma
3. Can use mobile phone to surf the Internet
4. Fluent in listening, speaking, reading and writing Chinese
5. Volunteer participation in this research

Exclusion Criteria:

1. Those who are unconscious or unable to communicate clearly
2. Those who have been diagnosed with mental illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline score of the Stoma Care Awareness Assessment at the first and second months after discharge | Data will be collected before discharge(baseline-T0), after discharge in the first(T1) and second(T2) months.
  The knowledge of self-care for their colostomy The Stoma Care Cognition Assessment Form is developed by researchers based on related literature on stoma care. There are 10 items, including normal/abnormal judgments of stoma, replacement of stoma, nutrition, and activities, all of which are single-choice questions. Each question is counted with 10 points, and the total score is 100 points. The higher the score, the better the respondent's awareness of stoma care.
Change from the baseline score of the General Anxiety Disorder-7(GAD-7) at the first and second months after discharge | Data will be collected before discharge(baseline-T0), after discharge in the first(T1) and second(T2) months.
  The GAD-7 (Spitzer et al., 2006) is a one-dimensional instrument designed to detect generalized anxiety disorder symptoms as defined in the DSM-IV. The item scores range from 0 (not at all) to 3 (nearly every day), resulting in a sum score range from 0 to 21. The higher scores reflect greater anxiety severity.
Change from the baseline score of the Patient Health Questionnaire-9(PHQ-9) at the first and second months after discharge | Data will be collected before discharge(baseline-T0), after discharge in the first(T1) and second(T2) months.
  The nine items of the PHQ-9 are designed to capture the nine Diagnostic and Statistical Manual of Mental Disorders (DSM) symptom criteria for a major depressive episode. Response options on the items range from "not at all" (0 points) to "nearly every day"(3 points). As a severity measure, the PHQ-9 score can range from 0 to 27.
Change from the baseline score of the WHO Quality of Life-BREF,WHOQOL- BREF at the first and second months after discharge | Data will be collected before discharge(baseline-T0), after discharge in the first(T1) and second(T2) months.
  The Taiwan version of the WHOQOL-BREF questionnaire is based on the WHOQOL-BREF. The 26 questions of the WHOQOL-BREF are kept and translated into Chinese. In addition, two local questions are added to make a total of 28 questions. Divided into four categories, one is the physiological category (including physiology and independence), with a total of 7 questions; the second is the psychological category (including psychology, soul, religion, and personal beliefs), with a total of 6 questions; the third is the social relationship category, with a total of 4 questions; The fourth is the environmental project, a total of 9 questions; the other 2 questions are the overall assessment questions. Each question in the questionnaire is scored using Likert's five-point scale. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
The User Version of the Mobile Application Rating Scale: uMARS | Data will be collected after discharge in the second month(T2).
  The mobile app score scale is a tool developed by Stoyanov et al. (2015) to classify and evaluate the quality of health-related mobile device apps. The scale has 23 questions and uses a 5-point scoring method (1-no Adequate, 2-Poor, 3-Acceptable, 4-Good, 5-Excellent). In addition, in order to adapt to the different situations of each mobile device application, there is also an option of "not applicable" for each question. Divided into four objective quality dimensions-participation (5 questions), functionality (4 questions), aesthetics (3 questions) and information quality (7 questions), and a subjective quality dimension (4 questions) contains to will it be recommended, frequency of use in the future, willingness to pay for it, and overall rating. The score calculation method is based on the average of the scores of each quality dimension and the total scale, the highest is 5 points, and the lowest is 1 point. The higher the average score, the better the quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Hung, BS, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dabas H, Sharma KK, Joshi P, Agarwala S. Video teaching program on management of colostomy: Evaluation of its impact on caregivers. J Indian Assoc Pediatr Surg. 2016 Apr-Jun;21(2):54-6. doi: 10.4103/0971-9261.176933. PMID 27046974
- [Background] Kim H, Goldsmith JV, Sengupta S, Mahmood A, Powell MP, Bhatt J, Chang CF, Bhuyan SS. Mobile Health Application and e-Health Literacy: Opportunities and Concerns for Cancer Patients and Caregivers. J Cancer Educ. 2019 Feb;34(1):3-8. doi: 10.1007/s13187-017-1293-5. PMID 29139070
- [Background] Putranto D, Rochmawati E. Mobile applications for managing symptoms of patients with cancer at home: A scoping review. Int J Nurs Pract. 2020 Aug;26(4):e12842. doi: 10.1111/ijn.12842. Epub 2020 Apr 29. PMID 32347599
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964
- [Background] Sun V, Ercolano E, McCorkle R, Grant M, Wendel CS, Tallman NJ, Passero F, Raza S, Cidav Z, Holcomb M, Weinstein RS, Hornbrook MC, Krouse RS. Ostomy telehealth for cancer survivors: Design of the Ostomy Self-management Training (OSMT) randomized trial. Contemp Clin Trials. 2018 Jan;64:167-172. doi: 10.1016/j.cct.2017.10.008. Epub 2017 Oct 16. PMID 29051047